CLINICAL TRIAL: NCT03197974
Title: Web-based Intervention With Email Support to Improve Quality of Life in Late Stage Bipolar Disorder (ORBIT): Randomised Controlled Trial
Brief Title: RCT of a Web-based Intervention to Improve Quality of Life in Late Stage Bipolar Disorder (ORBIT)
Acronym: ORBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: University of British Columbia (Other); National Health and Medical Research Council, Australia (Other); University of California, Berkeley (Other); Lancaster University (Other); Deakin University (Other); Australian National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ORBIT; APP1102097 (Other Grant/Funding Number: National Health and Medical Research Council Australia)
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder, Currently in Remission
Keywords: stage; online; self-help; coaching support; quality of life; mindfulness; psychoeducation; persuasive systems design; psychosocial
MeSH Terms: conditions — Bipolar Disorder | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: It is a prospective, parallel group, rater-blind, superiority RCT with a 1:1 allocation ratio comparing two websites designed to improve QoL in late stage bipolar disorder. Follow-up time points are immediate post-treatment (primary outcome timepoint), 3-month and 6-month follow-ups. To minimise the risk of bias, we are not publicising which arm is expected to be superior in terms of the primary outcome. Note that we expect that both arms will lead to QoL benefits, and the statistical analysis plan is agnostic about the superiority of the experimental intervention over active control on a number of secondary outcome variables. In both arms, usual management will continue throughout, with medication and psychosocial intervention changes monitored at follow-up interviews. The study setting is online, and participation in both arms will be through a secure server at Swinburne University's National eTherapy Centre (NetC).
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessors will be blinded as to treatment allocation. To maintain blinding, the Assessor will not be involved in intervention delivery and participants will be instructed not to discuss treatment with their interviewer. When an interview leads to unblinding, the assessor will be replaced.
  Participants will be blinded as to the primary hypothesis of which website will have superior benefits for QoL, but will of course be aware of the intervention they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness for Bipolar (Other): Introduction to, and training in the skills of mindfulness, self-compassion, and values-oriented action, and how these can be applied to managing symptoms of bipolar disorder.
  Interventions: Behavioral: Mindfulness for Bipolar
- Psychoeducation for Bipolar (Other): Information about bipolar disorder and the patient's role in managing the condition, including identifying triggers, and responding to early warning signs of episodes, and developing a healthy lifestyle
  Interventions: Behavioral: Psychoeducation for Bipolar

INTERVENTIONS:
Behavioral: Mindfulness for Bipolar — Brief online self-management program with email coaching support
  Arms: Mindfulness for Bipolar
Behavioral: Psychoeducation for Bipolar — Brief online self-management program with email coaching support
  Arms: Psychoeducation for Bipolar

SUMMARY:
The aim of this study is to improve outcomes in people with bipolar disorder (BD) by comparing two new online interventions specifically designed to improve quality of life amongst people who have had multiple (10 or more) episodes of BD.

DETAILED DESCRIPTION:
People who have had significant experience with bipolar disorder (defined here as 10 or more episodes) may not benefit from existing psychosocial interventions targeting symptoms and relapse, and may be better served by interventions targeting quality of life (QoL). Our international team of researchers, clinicians and consumers has developed two different online interventions, both of which there is reason to believe will be useful. Both interventions are brief, with 4 weeks of new online content released weekly, plus one additional week of application. This 5-week 'active phase' is supported by email contact with a personal online coach. The remainder of the 6 months of participant involvement in the trial includes continued access to the website (without coaching support) and follow-up assessments. Both arms are equivalent in using cutting-edge internet technologies and design features to help people engage with the therapeutic content and generalise it into their real lives. The websites have been developed following best-practice principles of persuasive system design, and rely heavily on consumer videos, social engagement through discussion boards, personalised feedback, and intuitive content structure to maximise engagement.

Australia's NHMRC has funded a 4-year project (2016-2019) to develop and compare the effectiveness of the two websites in terms of a range of outcomes, primarily QoL. The randomized controlled trial (RCT) will definitively assess the QoL benefits of two websites for late stage Bipolar Disorder. The RCT has been designed to optimise various aims: minimise risk of bias to support definitive scientific findings (internal validity), support ready dissemination should outcomes be positive (external validity, end-user involvement), and to optimally manage the risks inherent in the population being studied. We expect to find definitive evidence of the comparative QoL benefits of the two interventions, and insights about secondary outcomes including self-rated state anxiety, self-rated depression, and clinician-rated depression. A number of clinical and functional secondary outcomes will also be explored, as will hypothesised mediators and baseline moderators of QoL outcomes. Economic analysis based on cost-consequence analysis, and a range of process evaluations will also be conducted.

A total of 300 participants will be block randomised to provide power to identify a small-moderate treatment effect on QoL. Participants will be blinded as to the experimental intervention. The study uses a single-site (internet-based) design, with advertising occurring primarily online, but also through traditional methods via clinical networks of the researchers in Australia, United Kingdom (UK), Canada and the US. Major assessment time points are baseline, post-treatment (primary endpoint), 3 months post-baseline and 6 months post-baseline. Participants will be remunerated for assessments, which include both online questionnaires and a (blinded) semi-structured clinical interview by phone.

A multi-layered risk-management approach has been developed based on our experience with online interventions for bipolar disorder and psychosis. First and foremost, we explain to participants that their participation does not replace usual care, and no emergency assistance is available through the website (a link to the international site unsuicide is provided). This devolving of responsibility to the participant is reinforced by the inclusion criterion of being under the care of a medical practitioner and having access to local emergency services. Second, both intervention sites contain general information about the potential risks (e.g., generating distress) of the interventions, as well as specific alerts to the potential challenges of particular exercises. Third, a comprehensive 'red flag decision tree' has been developed to guide the team's response to any risk issues arising (see Table 2). Finally, any adverse events arising will be reviewed weekly in the trial executive committee.

ELIGIBILITY:
To ensure ready translation, minimally restrictive inclusion and exclusion criteria will be set.

Inclusion Criteria:

* diagnosis of BD from a mental health professional
* diagnosis of BD (BD I, BD II or Other Specified Bipolar and Related Disorder) confirmed by semi-structured interview using DSM-5 (Diagnostic and statistical manual of mental disorders-5) criteria, excluding criteria that mania/hypomania require abnormalities of activity/energy.
* must have experienced 10 or more episodes of mania, hypomania or depression
* must be under the care of and able to provide phone/mail contact details for a nominated medical practitioner
* must have local access to emergency services
* must have sufficient understanding of written and spoken English
* must have ready daily access to the internet and adequate internet literacy
* aged between 18 - 65 years

Exclusion criteria:

* currently experiencing an episode of depression or hypo/mania
* currently psychotic or actively suicidal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Brief QoL.BD | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  Self-report measure to assess quality of life.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Scale (MADRS) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A clinician-rated scale to assess depression symptoms.
Change in Young Mania Rating Scale (YMRS) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A clinician-rated scale to assess manic symptoms.
Change in Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of depression.
Change in Depression Anxiety Stress Scale (DASS-21, Anxiety and Stress Scales only) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of anxiety and stress symptoms.
Change in Functional Assessment Staging Test (FAST) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A clinician-rated scale to assess functioning across 6 different domains.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of sleep quality.
Change in Sleep, Circadian Rhythms and Mood questionnaire (SCRAM) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess overlap between sleep, circadian rhythms and mood.
Occurrence of intervention-related relapse | Immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  Using the Time to Intervention for Mood Episode (TIME) and a modified version of the MINI International Neuropsychiatric Interview (MINI) to determine treatment-related relapse events.

OTHER OUTCOMES:
Change in Resource Use Questionnaire | Baseline, 3 and 6 months.
  A self-report measure of health service use.
Change in Assessment of Quality of Life 8dimension (AQol8d) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of quality of life.
Change in Five Facet Mindfulness Questionnaire (FMQ) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of mindfulness.
Change in Self-Compassion Scale (SCS) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of self-compassion.
Change in Difficulties in Emotion Regulation Scale-16 Item (DERS-16) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess multiple aspects of emotion dysregulation.
Change in Ruminative Responses Scale (section of the Response Styles Questionnaire) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure of tendency to ruminate.
Change in Responses to Positive Affect scale (RPA) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess rumination and dampening.
Change in Non-attachment to Ego Scale | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess non-attachment to self.
Change in Depressive Experience Questionnaire Self-Criticism Six-Item Scale (DEQ-SC6) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess self-criticism.
Change in the Short revised almost perfect scale (SAPS) | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  A self-report measure to assess perfectionism.
Change in adherence to medication. | Baseline, immediately post-intervention (post the 5 week active phase), 3 and 6 months.
  Self-reported adherence to medication.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Murray, Principal Investigator — Swinburne University of Technology
Locations (1):
- Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fletcher K, Foley F, Thomas N, Michalak E, Berk L, Berk M, Bowe S, Cotton S, Engel L, Johnson SL, Jones S, Kyrios M, Lapsley S, Mihalopoulos C, Perich T, Murray G. Web-based intervention to improve quality of life in late stage bipolar disorder (ORBIT): randomised controlled trial protocol. BMC Psychiatry. 2018 Jul 13;18(1):221. doi: 10.1186/s12888-018-1805-9. PMID 30001704